CLINICAL TRIAL: NCT00004261
Title: A Phase I Trial of the Hypoxia Detection Agent EF5 (NSC 684681) in Patients With Cervix and Breast and Prostate Carcinomas, and High Grade Soft Tissue Sarcomas
Brief Title: EF5 Prior to Surgery or Biopsy in Patients With Breast, Prostate, or Cervical Cancer or High Grade Soft Tissue Sarcoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of patient accrual
Sponsor: University Health Network, Toronto (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Diagnostic
Other Study IDs: CAN-OCI-T98-0048; CDR0000067516 (Registry Identifier: PDQ (Physician Data Query)); NCI-T98-0048
Record Dates: First submitted 2000-01-28; First posted 2003-12-11 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Breast Cancer; Cervical Cancer; Head and Neck Cancer; Prostate Cancer; Sarcoma
Keywords: stage I breast cancer; stage II breast cancer; stage IV breast cancer; stage IIIA breast cancer; breast cancer in situ; recurrent breast cancer; stage IIIB breast cancer; stage 0 cervical cancer; stage III cervical cancer; recurrent cervical cancer; stage IB cervical cancer; stage IIB cervical cancer; stage IVB cervical cancer; stage IA cervical cancer; stage IIA cervical cancer; stage IVA cervical cancer; inflammatory breast cancer; stage III adult soft tissue sarcoma; recurrent adult soft tissue sarcoma; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage IV prostate cancer; recurrent prostate cancer; stage I nasopharyngeal cancer; stage II nasopharyngeal cancer; stage III nasopharyngeal cancer; stage IV nasopharyngeal cancer; recurrent nasopharyngeal cancer; stage 0 paranasal sinus and nasal cavity cancer; stage 0 nasopharyngeal cancer; stage 0 oropharyngeal cancer; stage 0 laryngeal cancer; stage 0 hypopharyngeal cancer; stage I salivary gland cancer; stage II salivary gland cancer; stage III salivary gland cancer; stage IV salivary gland cancer; recurrent salivary gland cancer; untreated metastatic squamous neck cancer with occult primary; recurrent metastatic squamous neck cancer with occult primary; stage 0 lip and oral cavity cancer; stage IV adult soft tissue sarcoma; stage I lip and oral cavity cancer; stage II lip and oral cavity cancer; stage III lip and oral cavity cancer; stage IV lip and oral cavity cancer; recurrent lip and oral cavity cancer; stage I hypopharyngeal cancer; stage II hypopharyngeal cancer; stage III hypopharyngeal cancer; stage IV hypopharyngeal cancer; recurrent hypopharyngeal cancer; stage I laryngeal cancer; stage II laryngeal cancer; stage III laryngeal cancer; stage IV laryngeal cancer; recurrent laryngeal cancer; stage I paranasal sinus and nasal cavity cancer; stage II paranasal sinus and nasal cavity cancer; stage III paranasal sinus and nasal cavity cancer; stage IV paranasal sinus and nasal cavity cancer; recurrent paranasal sinus and nasal cavity cancer; stage I oropharyngeal cancer; stage II oropharyngeal cancer; stage III oropharyngeal cancer; stage IV oropharyngeal cancer; recurrent oropharyngeal cancer; stage II adult soft tissue sarcoma; stage I adult soft tissue sarcoma
MeSH Terms: conditions — Breast Neoplasms; Uterine Cervical Neoplasms; Head and Neck Neoplasms; Prostatic Neoplasms; Sarcoma; Breast Carcinoma In Situ; Uterine Cervical Dysplasia; Inflammatory Breast Neoplasms; Nasopharyngeal Neoplasms; Oropharyngeal Neoplasms; Laryngeal Neoplasms; Hypopharyngeal Neoplasms; Salivary Gland Neoplasms; Mouth Neoplasms | interventions — Flow Cytometry; Fluorescent Antibody Technique; Immunohistochemistry; Biopsy

INTERVENTIONS:
Drug: EF5
Other: flow cytometry
Other: fluorescent antibody technique
Other: immunohistochemistry staining method
Procedure: biopsy

SUMMARY:
RATIONALE: EF5 may detect the presence of oxygen in tumor cells and help plan effective cancer treatment.

PURPOSE: Phase I trial to study the effectiveness of EF5 in detecting the presence of oxygen in tumor cells of patients who are undergoing surgery or biopsy for breast, prostate, or cervical cancer or high grade soft tissue sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the optimal dose of etanidazole derivative EF5 that is safely tolerated and provides optimal binding in resected tumor specimens or tumor biopsies in patients with breast, head and neck, prostate, or cervical carcinoma or high grade soft tissue sarcomas. II. Define the toxic effects of EF5 in this patient population.

OUTLINE: This is a dose-escalation study. Patients receive etanidazole derivative EF5 IV over 1-2 hours. Approximately 24-48 hours after EF5 treatment, patients undergo surgical resection or biopsy of tumor. Cohorts of 6 patients receive escalating doses of EF5 until the maximum tolerated dose (MTD) or optimal dose is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. The optimal dose is defined as the dose level at or preceding the MTD and resulting in optimal tumor-to-normal-tissue binding. Patients are followed at 28 days.

PROJECTED ACCRUAL: A total of 18-36 patients will be accrued for this study within 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven breast, head and neck, prostate, or cervical carcinoma or high grade (defined as grades 2 or 3) soft tissue sarcoma Sarcoma tumors must be confined to truncal or extremity locations Must have a clinical condition and physiologic status which demonstrates that the appropriate or standard initial therapy for the tumor is surgical biopsy or resection Tumors no greater than 15 cm in any diameter Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 18 and over Menopausal status: Not specified Performance status: ECOG 0 or 1 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count greater than 2,000/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin less than 2.0 mg/dL Renal: Creatinine less than 2.0 mg/dL OR Creatinine clearance greater than 50 mL/min Cardiovascular: No significant cardiac disease that would preclude the safe use of general anesthesia Pulmonary: No significant pulmonary disease that would preclude the safe use of general anesthesia Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for 1 month after study No grade 3 or 4 peripheral neuropathy

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Not specified Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-12; Primary Completion 2002-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Fyles, MD, Study Chair — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada